CLINICAL TRIAL: NCT02957877
Title: Low-molecular Heparin Infusion as Anticoagulation for Nocturnal Home Hemodialysis
Brief Title: LMWH Infusion as Anticoagulation for Home HD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alice Ho Miu Ling Nethersole Hospital (Other)
Responsible Party: Principal Investigator, Steve Siu-Man Wong, Associate Consultant, Alice Ho Miu Ling Nethersole Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015.415
Record Dates: First submitted 2016-11-02; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Endstage Renal Disease
Keywords: Anticoagulation; Anti-Xa activity; Low-molecular weight heparin; Unfractionated heparin
MeSH Terms: interventions — Nadroparin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LMWH arm (Experimental): 8-hour hemodialysis is performed on alternate day for a week at the dialysis unit (i.e. 3 sessions) by using low-molecular weight heparin (nadroparin) as anticoagulation
  Interventions: Drug: Nadroparin
- UFH arm (Active Comparator): 8-hour hemodialysis is performed on alternate day for a week at the dialysis unit (i.e. 3 sessions) by using unfractionated heparin as anticoagulation
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: Nadroparin — A nadroparin infusion regimen (loading dose of 35 IU/kg, followed by 10 IU/kg per hour for 6 hours) is administered as anticoagulation during the 8-hour hemodialysis.
  Other Names: Fraxiparine
  Arms: LMWH arm
Drug: Unfractionated heparin — The individualized unfractionated heparin infusion regimen currently employed by the recruited patients in their home dialysis treatment is administered as anticoagulation during the 8-hour hemodialysis.
  Arms: UFH arm

SUMMARY:
There is a lack of data in the literature about the use of low-molecular weight heparin (LMWH) as anticoagulation for nocturnal home hemodialysis (NHHD). This study aims to evaluate the efficacy and safety of LMWH, administered by infusion method, as compared to unfractionated heparin as anticoagulation for NHHD treatment.

DETAILED DESCRIPTION:
Low-molecular weight heparin (LMWH) and unfractionated heparin (UFH) are established systemic anticoagulants for the patients who receive conventional thrice-weekly hemodialysis in absence of significant bleeding risk. For the patients who undergo nocturnal home hemodialysis (NHHD), LMWH is seldom utilized because of the need of an additional bolus injection during a long dialysis treatment, which is impractical as the patients are sleeping during hemodialysis. Moreover, there is a potential risk of LMWH accumulation due to its longer half-life. As there is a paucity of data in the literature on the use of LMWH for NHHD treatment, this trial is conducted to assess the safety and efficacy of LMWH, administered by infusion method, in this particular group of dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent NHHD patients who have received >1 year dialysis with unfractionated heparin as anticoagulant
* Age >= 18
* Informed consent available

Exclusion Criteria:

* History of intolerance to LMWHs during HD
* Receiving warfarin or other oral anticoagulant
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Prothrombin time | Pre-dialysis; the 2nd, 4th, 6th and 8th hours of dialysis
  Prothrombin time is monitored in both of the LMWH and UFH arms
Activated partial thromboplastin time | Pre-dialysis; the 2nd, 4th, 6th and 8th hours of dialysis
  Activated partial thromboplastin time is monitored in both of the LMWH and UFH arms
Anti-Xa level | Pre-dialysis; the 2nd, 4th, 6th and 8th hours of dialysis; 24 hours after administration of LMWH
  Anti-Xa level is only monitored in the LMWH arm
Dialyser urea and creatinine clearances | At 15 mins after starting hemodialysis and 15 mins before the end of hemodialysis
  Dialyser urea and creatinine clearances are evaluated in both of the LMWH and UFH arms
Dialyser thrombus score | At the end of hemodialysis (8th hour)
  Dialyser thrombus score is evaluated in both of the LMWH and UFH arms

CONTACTS AND LOCATIONS:
Overall Officials: Steve Siu-Man Wong, MBChB, FRCPC, Principal Investigator — Alice Ho Miu Ling Nethersole Hospital
Locations (1):
- Alice Ho Miu Ling Nethersole Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593